CLINICAL TRIAL: NCT04644965
Title: Evaluation of the Motor Activity, Cardiopulmonary Performance Capacity and Quality of Life in Patients Born With a Congenital Abdominal Wall Defect
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 32-231 ex 19/20
Record Dates: First submitted 2020-11-19; First posted 2020-11-25 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-01

CONDITIONS: Abdominal Wall Defect
MeSH Terms: interventions — Ultrasonography; Gait Analysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Abdominal Wall Defect: patients born with an abdominal wall defect
  Interventions: Diagnostic Test: CombynTM Function & Spaces ECG; Diagnostic Test: Blood Taking; Diagnostic Test: Spiroergometry; Diagnostic Test: Dordel Koch Test (DKT); Diagnostic Test: Ultrasound; Diagnostic Test: Stance and gait analyses
- Control Group: age and sex matched Control Group
  Interventions: Diagnostic Test: CombynTM Function & Spaces ECG; Diagnostic Test: Blood Taking; Diagnostic Test: Spiroergometry; Diagnostic Test: Dordel Koch Test (DKT); Diagnostic Test: Ultrasound; Diagnostic Test: Stance and gait analyses

INTERVENTIONS:
Diagnostic Test: CombynTM Function & Spaces ECG — Multi-frequency impedance measurement to assess the muscle and fat mass
Diagnostic Test: Blood Taking — Sampling of blood of the finger pad to assess liver function
Diagnostic Test: Spiroergometry — Spiroergometry to assess cardiopulmonary capacity. The intensity will be raised in steps until total exhaustion. In between each step we will take blood of the ear lobe to determine the lactate level
Diagnostic Test: Dordel Koch Test (DKT) — Dordel Koch Test (DKT) to evaluate the motor activity. The DKT is a heterogeneous test battery for children and adolescents and consists of seven parts: lateral jumping, sit and reach, situps, long stand jump, one-legged stand, push-ups and 6-min-run
Diagnostic Test: Ultrasound — Ultrasound for abdominal wall muscles
Diagnostic Test: Stance and gait analyses — Stance and gait analyses for measuring the core stability

SUMMARY:
The two most common congenital abdominal wall defects (AWD) are gastroschisis and omphalocele. Prenatal detection is often possible and the defects are differentiated by the presence or absence of a sac around the eviscerated organs. A omphalocele occurs in 0.6-4.8 in 10,000 live births compared to 4.5 in 10,000 live births with gastroschisis. In the last years a rising incidence of gastroschisis has been shown worldwide.

Both forms of AWDs necessitate early surgical intervention, mostly in one or two stages, and support at an intensive care unit in the first days of life. Additionally, patients need parenteral feeding in the first weeks of life. The outcome depends on the size of the defect and on the associated malformations.

The literature about long-term outcome of these malformations is scarce. Some publications have reported long-term complications like redo-surgical procedures because of fascial gaps or umbilical or incisional hernias. Furthermore, stool irregularities, abdominal pain and several admission to the hospital due to ileus or sub-ileus have been described. Additionally, half of the patients are unsatisfied with the cosmetic result.

Some other studies have shown that children born with an AWD have the same quality of life (QoL) compared with the healthy community.

Nevertheless, patients with AWDs need a standardized, structured and multimodal long-time follow-up program to be able to detect any problems early and give advice to understand their illness in order to achieve the same QoL as healthy children.

Therefore, the aim of this dissertation will be:

* to prospectively assess the motor activity, cardiopulmonary performance capacity and QoL of patients treated with AWDs in our Department
* to suggest a new standardized follow-up protocol for patients born with an AWD

ELIGIBILITY:
Inclusion Criteria:

* All patients born with an abdominal wall defect

Exclusion Criteria:

* mental disease

Ages: 6 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: All patients born with an abdominal wall defect between 6-18years old are invited personally for examinations.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Motor Activity | 30 minutes
  Comparison of the Dordel Koch Test between the two groups. (T-Test or Mann-Withney-U)
Cardiopulmonary Performance Capacity - lung function | 30 minutes
  Comparing relative lung function [%] between the two groups.(T-Test or Mann-Withney-U)
Cardiopulmonary Performance Capacity - peak VO2 | 30 minutes
  Comparing peak VO2 between the two groups.(T-Test or Mann-Withney-U)
Gastrointestinal Quality of Life | 15 minutes
  Gastrointestinal Quality of Life Index (GIQLI): most desirable option: 4 points, least desirable option: 0 points GIQLI score: sum of the points - Score Range: 0-148 Compare the mean between the two groups (T-Test or Mann-Withney-U)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Frybova B, Kokesova A, Zemkova D, Mixa V, Vlk R, Rygl M. Quality of life in patients with gastroschisis is comparable with the general population: A questionnaire survey. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2017 Mar;161(1):75-79. doi: 10.5507/bp.2016.059. Epub 2016 Dec 13. PMID 27982137
- [Background] Snoep MC, de Heus R, Manten GTR, Lap CCMM, Snoeker BAM, Lindeboom MYA. Gastro-intestinal function and quality of life are favorable in adolescent and adult gastroschisis patients. Early Hum Dev. 2020 Feb;141:104936. doi: 10.1016/j.earlhumdev.2019.104936. Epub 2019 Dec 23. PMID 31874371
- [Background] Harris EL, Minutillo C, Hart S, Warner TM, Ravikumara M, Nathan EA, Dickinson JE. The long term physical consequences of gastroschisis. J Pediatr Surg. 2014 Oct;49(10):1466-70. doi: 10.1016/j.jpedsurg.2014.03.008. PMID 25280647
- [Background] Kaiser MM, Kahl F, von Schwabe C, Halsband H. [Omphalocele and gastroschisis. Outcome--complications--follow-up--quality of life]. Chirurg. 2000 Oct;71(10):1256-62. doi: 10.1007/s001040051212. German. PMID 11077588